CLINICAL TRIAL: NCT04960150
Title: EFFECTS OF ACUPUNCTURE ON LEG MUSCLE STRENGTH: RANDOMIZED CONTROLLED TRIAL IN SPORTS STUDENTS
Brief Title: EFFECTS OF ACUPUNCTURE ON LEG MUSCLE STRENGTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Wahyuningsih Djaali, Lecturer, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-05-0541
Record Dates: First submitted 2021-06-23; First posted 2021-07-13 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Health, Subjective; Muscle Strength
Keywords: acupuncture; press tack needle; leg strength

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Intervention of press tack needle acupuncture
  Interventions: Device: Press tack needle
- Control group (Placebo Comparator): Intervention of placebo acupuncture
  Interventions: Device: Plesterin

INTERVENTIONS:
Device: Press tack needle — Press tack needle acupuncture using "Seirin Pyonex" sized 0.20x1.2mm
  Arms: Acupuncture group
Device: Plesterin — Plesterin
  Arms: Control group

SUMMARY:
Press tack needle is one of the acupuncture modalities in the form of needles that are attached to the skin, and can be left attached to the skin for several days which makes its use much easier than conventional acupuncture.

The purpose of this study was to determine how the effect of press tack needle acupuncture on leg muscle strength performed on sports students.

Research subjects as many as 30 people were randomized into two groups, namely the intervention group and the control group. In the intervention group, acupuncture treatment was performed with a press tack needle at acupuncture points on the legs. The leg muscle strength was measured using a leg dynamometer before and after the acupuncture intervention. Analyzed the difference in mean leg muscle strength before and after the intervention, and between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* willingness to fill out an informed consent form;
* age between 18-25 years;
* male;
* has a BMI value of 18.5-22.9 kg/m2;
* there is no history of injury or history of surgery on the lower extremities in the last three months;
* the individual is in good health.

Exclusion Criteria:

* absence or refusal to be examined and not cooperative.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Leg muscle strength | baseline (Before intervention)
  Measurement of leg muscle strength before the intervention, and compared between the two groups
Leg muscle strength | 35 minutes after intervention
  Measurement of leg muscle strength after the intervention, and compared between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Sport Science Faculty, Universitas Negeri Jakarta, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No